CLINICAL TRIAL: NCT06389162
Title: The Influence of Dorsolateral Prefrontal Cortex Transcranial Direct Current Stimulation on Muscle Fatigue
Brief Title: Dorsolateral Prefrontal Cortex Transcranial Direct Current and Muscle Fatigue Stimulation on Muscle Fatigue
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Brach Poston, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UNLV-2024-115
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (Experimental): Transcranial direct current stimulation applied to the left dorsolateral prefrontal cortex
  Interventions: Device: transcranial direct current stimulation
- SHAM (Sham Comparator): SHAM transcranial direct current stimulation applied to the left dorsolateral prefrontal cortex
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation is a type of non-invasive brain stimulation that involves passing a weak current between two electrodes placed on the scalp.

SUMMARY:
The goal of this clinical trial is to learn if transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex (DLPFC) can impact muscle fatigue. The main questions it aims to answer are:

1. Does tDCS of the left DLPFC increase the time that a fatiguing contraction can be maintained?
2. Does tDCS of the left DLPFC decrease the rate of increase of muscle activity, force error, and standard deviation of force during a fatiguing contraction.

Researchers will compare tDCS of the left DLPFC to a SHAM stimulation (a type of stimulation that feels like real tDCS but does not elicit physiological effects) to see if tDCS of the left DLPFC works to reduce the progression of muscle fatigue.

Participants will:

Performing two experimental sessions held 3-10 days apart (usually 7 days) Perform a 9 hole pegboard test, maximum voluntary contractions, and a fatiguing contraction.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) delivered to the dorsolateral prefrontal cortex (DLPFC) can increase endurance time in lower body tasks. Therefore, the purpose of this study is to examine the effect of DLPFC-tDCS on the time to task failure (TTF) of a fatiguing contraction performed by hand muscles. The study will use a double-blind, randomized, SHAM-controlled, crossover design with each participant performing two experimental sessions held 3-7 days apart. The only difference between the two sessions will be the type of stimulation (tDCS or SHAM; counterbalanced) applied concurrent with the fatiguing contraction. The fatiguing contraction will involve gripping a manipulandum with the index finger and thumb. This will be accomplished by using a precision grip and matching an isometric target equal to 15% of the maximum voluntary contraction (MVC) for as long as possible until task failure.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Free from any neurological or psychiatric condition
3. Age between 18-50 years old
4. Right-handed (as determined by the Edinburgh Handedness Inventory)

Exclusion Criteria:

1. An uncontrolled medical condition (i.e. hypertension, diabetes, etc)
2. Metal in the skull or the eye, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain, cochlear implants, and metal fragments in the eye.
3. Hearing loss diagnosed by a doctor and requiring a hearing aid. Have had a brain tumor, a stroke, head trauma, epilepsy or a history of seizures, have a neurological disorder, a movement disorder, or have a head injury that involved being passed out for more than a few seconds.
4. History of migraines
5. implanted defibrillator or implanted neurostimulator
6. pregnant or thought to be pregnant. This must be an exclusion criterion as there are few medical papers available regarding the effects of tDCS on the unborn child/fetus or expectant mother. Thus, if you are pregnant or thought to be pregnant you cannot participate in the study. If you find out you are pregnant in the week timeframe between experiment 1 and experiment 2, you should withdraw from the study as we cannot perform the second experiment in that case.
7. Not done a similar fatigue study in the laboratory in the last 7 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to Task Failure | 5 months
  The time in seconds that a fatiguing contraction can be held
Fatigue Index | 5 months
  The percent decline in force between the maximum voluntary contractions performed before and after the fatiguing contraction

SECONDARY OUTCOMES:
Average EMG activity | 5 months
  The average EMG activity of the first dorsal interosseus muscle during the fatiguing contraction.
Force error | 5 months
  The average force error during the fatiguing contraction.
Standard deviation of force | 5 months
  The average standard deviation of force during the fatiguing contraction.
9 Hole Pegboard Test | 5 months
  9 Hole Pegboard Test time before and after the fatiguing contraction

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided